CLINICAL TRIAL: NCT06256263
Title: Linear Stapler Versus Conventional Repair of the Pharynx After Total Laryngectomy: Functional and Oncological Outcomes
Brief Title: Stapler Versus Conventional Pharyngeal Repair After Total Larygectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD.21.06.491
Record Dates: First submitted 2024-02-03; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Malignant Tumor of the Larynx
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stapler repair group (Active Comparator): pharyngeal repair after total laryngectomy was done by using a linear stapler
  Interventions: Procedure: total laryngectomy
- conventional repair group (Active Comparator): pharyngeal repair after total laryngectomy was done by the conventional method (stitching).
  Interventions: Procedure: total laryngectomy

INTERVENTIONS:
Procedure: total laryngectomy — pharyngeal repair after total laryngectomy

SUMMARY:
This study was done to investigate the efficacy and safety of the linear stapler closure of the pharynx after total laryngectomy.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing total laryngectomy for advanced laryngeal carcinoma in the study duration .

Exclusion Criteria:

* Infiltration of the safety margins proved by postoperative histopathology .
* Patients with tumor extension to the tongue base, or the hypopharynx .
* Patients who are unfit for surgery .
* Patients refusal to surgical treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of pharyngocutaneous fistula after total laryngectomy | four weeks
  to assess the effectiveness of pharyngeal repair and healing without pharyngocutaneous fistula

SECONDARY OUTCOMES:
assessment of the swallowing function after surgery | 6 months
  swallowing was evaluated subjectively by applying the Sydney Swallow Questionnaire, (SSQ) and was evaluated objectively by performing modified barium swallow and functional endoscopic evaluation of swallowing (FEES)

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University faculty of Medicine, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sansa-Perna A, Casasayas-Plass M, Rovira-Martinez C, Lopez-Vilas M, Garcia-Lorenzo J, Quer-Agusti M, Leon-Vintro X. Pharyngeal closure after a total laryngectomy: mechanical versus manual technique. J Laryngol Otol. 2020 Jul;134(7):626-631. doi: 10.1017/S0022215120001371. Epub 2020 Jul 29. PMID 32723416
- [Background] Sannikorn P, Pornniwes N. Comparison of outcomes for staple and conventional closure of the pharynx following total laryngectomy. J Med Assoc Thai. 2013 Mar;96 Suppl 3:S89-93. PMID 23682529
- [Background] Shan H, Gao Y, Liu L, Li M, Gao X, Li Y, Wang X, Ouyang D, Guo Z. Magnifying endoscopy with narrow-band imaging to assist the linear stapler closure of the pharynx during total laryngectomy. Am J Otolaryngol. 2018 Sep-Oct;39(5):511-514. doi: 10.1016/j.amjoto.2018.05.014. Epub 2018 May 28. PMID 29903625